CLINICAL TRIAL: NCT02896855
Title: A Phase III, Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Efficacy and Safety of Pertuzumab+Herceptin+Docetaxel Versus Placebo+Herceptin+Docetaxel in Previously Untreated HER2-Positive Metastatic Breast Cancer
Brief Title: A Study to Evaluate the Efficacy and Safety of Pertuzumab + Trastuzumab + Docetaxel Versus Placebo + Trastuzumab + Docetaxel in Previously Untreated Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Metastatic Breast Cancer
Acronym: PUFFIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YO29296
Record Dates: First submitted 2016-09-07; First posted 2016-09-12 (Estimated); Results first posted 2019-07-10 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; pertuzumab; Trastuzumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A: Placebo + Trastuzumab + Docetaxel (Active Comparator): Placebo matched to pertuzumab, trastuzumab (8-milligrams per kilogram [mg/kg] loading dose for Cycle 1, followed by 6 mg/kg for subsequent cycles), and docetaxel (75-milligrams per square meter [mg/m^2]) were administered by intravenous (IV) infusion every 3 weeks until disease progression or unacceptable toxicity.
  Interventions: Drug: Docetaxel; Drug: Placebo; Drug: Trastuzumab
- Arm B: Pertuzumab + Trastuzumab + Docetaxel (Experimental): Pertuzumab (840-mg loading dose for Cycle 1, followed by 420 mg for subsequent cycles), trastuzumab (8-mg/kg loading dose for Cycle 1, followed by 6 mg/kg for subsequent cycles), and docetaxel (75-mg/m^2) were administered by IV infusion every 3 weeks until disease progression or unacceptable toxicity.
  Interventions: Drug: Docetaxel; Drug: Pertuzumab; Drug: Trastuzumab

INTERVENTIONS:
Drug: Docetaxel — Docetaxel (75-mg/m^2) was administered by IV infusion every 3 weeks until disease progression or unacceptable toxicity.
Drug: Pertuzumab — Pertuzumab (840-mg loading dose for Cycle 1, followed by 420 mg for subsequent cycles) was administered by IV infusion every 3 weeks until disease progression or unacceptable toxicity.
  Other Names: Perjeta
  Arms: Arm B: Pertuzumab + Trastuzumab + Docetaxel
Drug: Placebo — Placebo matched to pertuzumab was administered by IV infusion every 3 weeks until disease progression or unacceptable toxicity.
  Arms: Arm A: Placebo + Trastuzumab + Docetaxel
Drug: Trastuzumab — Trastuzumab (8-mg/kg loading dose for Cycle 1, followed by 6 mg/kg for subsequent cycles) was administered by IV infusion every 3 weeks until disease progression or unacceptable toxicity.
  Other Names: Herceptin

SUMMARY:
This Phase III, randomized, double-blind, placebo-controlled, multicenter clinical trial in China will evaluate the efficacy and safety of pertuzumab + trastuzumab + docetaxel compared with placebo + trastuzumab + docetaxel in participants with previously untreated HER2-positive metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the breast with locally recurrent or metastatic disease that is suitable for chemotherapy
* HER2-positive metastatic breast cancer (MBC)
* Left ventricular ejection fraction (LVEF) greater than or equal to (>=) 55 percent (%) at baseline (within 42 days of randomization)
* Eastern Cooperative Oncology Group Performance Status of 0 or 1
* Women of childbearing potential and men should agree to use an effective form of contraception and to continue its use for the duration of study treatment and for at least 7 months after the last dose of study treatment (trastuzumab and/or pertuzumab)

Exclusion Criteria:

* History of anti-cancer therapy for MBC (with the exception of one prior hormonal regimen for MBC)
* History of approved or investigative tyrosine kinase/HER inhibitors for breast cancer in any treatment setting, except trastuzumab used in the neoadjuvant or adjuvant setting
* History of systemic breast cancer treatment in the neo-adjuvant or adjuvant setting with a disease-free interval from completion of the systemic treatment (excluding hormonal therapy) to metastatic diagnosis of less than (<) 12 months
* History of persistent Grade >= 2 hematologic toxicity resulting from previous adjuvant therapy
* Grade >= 3 peripheral neuropathy at randomization
* History of other malignancy within the last 5 years, except for carcinoma in situ of the cervix or non-melanoma skin carcinoma that has been previously treated with curative intent
* Current clinical or radiographic evidence of central nervous system (CNS) metastases
* History of exposure to cumulative doses of anthracyclines
* Current uncontrolled hypertension or unstable angina
* History of congestive heart failure (CHF) of any New York Heart Association (NYHA) classification, or serious cardiac arrhythmia requiring treatment
* History of myocardial infarction within 6 months of randomization
* History of LVEF decrease to < 50% during or after prior trastuzumab neo-adjuvant or adjuvant therapy
* Current dyspnea at rest due to complications of advanced malignancy, or other diseases that require continuous oxygen therapy
* Inadequate organ function within 28 days prior to randomization
* Current severe, uncontrolled systemic disease
* Major surgical procedure or significant traumatic injury within 28 days prior to study treatment start or anticipation of the need for major surgery during the course of study treatment
* Pregnant or lactating women
* History of receiving any investigational treatment within 28 days of randomization
* Current known infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV), or active hepatitis B virus (HBV)
* Receipt of intravenous (IV) antibiotics for infection within 14 days of randomization
* Current chronic daily treatment with corticosteroids (excluding inhaled steroids)
* Known hypersensitivity to any of the protocol-specified study treatments
* Concurrent participation in an interventional or noninterventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2016-09-13 (Actual); Primary Completion 2018-06-27 (Actual); Study Completion 2021-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (15):
- China (15):
  - CHINESE ACADEMY OF MEDICAL SCIENCE; CANCER INST. & HOSPITAL; Medical ward, Beijing
  - Beijing Cancer Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - the First Hospital of Jilin University, Changchun
  - Changzhou First People's Hospital, Changzhou
  - West China Hospital, Sichuan University, Chengdu
  - The 900th Hospital of PLA joint service support force, Fuzhou
  - Guangdong General Hospital, Guangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Jiangsu province hospital; surgery on galactophore, Nanjing
  - Jiangsu Cancer Hospital, Nanjing
  - Fudan University Shanghai Cancer Center, Shanghai
  - First Hospital of China Medical University, Shenyang
  - Liaoning cancer Hospital & Institute, Shenyang
  - Zhejiang Cancer Hospital, Zhejiang

REFERENCES:
- [Derived] Xu B, Li W, Zhang Q, Shao Z, Li Q, Wang X, Li H, Sun T, Yin Y, Zheng H, Feng J, Zhang H, Lei G, Restuccia E. Pertuzumab, trastuzumab, and docetaxel for Chinese patients with previously untreated HER2-positive locally recurrent or metastatic breast cancer (PUFFIN): a phase III, randomized, double-blind, placebo-controlled study. Breast Cancer Res Treat. 2020 Aug;182(3):689-697. doi: 10.1007/s10549-020-05728-w. Epub 2020 Jun 20. PMID 32564260

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Placebo + Trastuzumab + Docetaxel: Placebo matched to pertuzumab, trastuzumab (8-milligrams per kilogram [mg/kg] loading dose for Cycle 1, followed by 6 mg/kg for subsequent cycles), and docetaxel (75-milligrams per square meter [mg/m^2]) were administered by intravenous (IV) infusion every 3 weeks until disease progression or unacceptable toxicity. Following the primary analysis and upon approval of protocol version 4 (07-March-2020), the treatment assignment of participants in Arm A who were still on study treatment was unblinded, allowing the investigators to present those participants with the option to cross over and receive pertuzumab (in place of placebo) in addition to trastuzumab and docetaxel.
Period: Overall Study
Arm/Group | Arm A: Placebo + Trastuzumab + Docetaxel | Arm B: Pertuzumab + Trastuzumab + Docetaxel
Started (Intent-to-Treat (ITT) Population) | 121 | 122
Received Any Study Treatment (Safety Population) | 120 | 122
Crossed Over From Placebo to Receive Pertuzumab | 12 (From 07-March-2020, 12 participants randomized to the Placebo arm crossed over to open-label pertuzumab.) | 0
Completed | 49 | 69
Not Completed | 72 | 53
Not completed — Death | 50 | 40
Not completed — Lost to Follow-up | 15 | 9
Not completed — Withdrawal by Subject | 7 | 4

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population: consists of all randomized participants, regardless of whether they received any study treatment. Participants are grouped according to the treatment group to which they were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Placebo + Trastuzumab + Docetaxel | Arm B: Pertuzumab + Trastuzumab + Docetaxel | Total
Number analyzed (Participants) | 121 | 122 | 243
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (11.2) | 50.7 (10.6) | 51.0 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 122 | 243
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 121 | 122 | 243
Disease Type: Visceral or Non-Visceral Disease [Count of Participants; unit: Participants]
  Visceral Disease | 86 | 88 | 174
  Non-Visceral Disease | 35 | 34 | 69
Hormone Receptor Status [Count of Participants; unit: Participants]
  Estrogen and Progesterone Receptor Negative | 48 | 53 | 101
  Estrogen and/or Progesterone Receptor Positive | 73 | 69 | 142
Measurable or Non-Measurable Disease, According to RECIST v1.1 [Count of Participants; unit: Participants]
  Measurable Disease | 97 | 105 | 202
  Non-Measurable Disease | 24 | 17 | 41

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival, as Determined by the Investigator Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: Progression-free survival (PFS) was defined as the time from randomization to first occurrence of progressive disease (PD), as determined by the investigator using RECIST v1.1, or death from any cause within 18 weeks after the last tumor assessment, whichever occurred first. As per RECIST v1.1, PD is defined as a 20% increase in the sum of the diameters of target lesions, an increase in size of measurable lesions by at least 5 millimeters (mm), and the appearance of new lesions. The Kaplan-Meier approach was used to estimate median PFS for each treatment arm. Data for participants who did not have a PFS event were censored at the time of the last tumor assessment (if no tumor assessments performed after baseline, at randomization plus 1 day).
Time Frame: From date of randomization until date of PFS event (Median [range] time on study for Arm A vs. Arm B at Primary analysis: 57.14 [3.3-93.3] weeks vs. 59.64 [0.9-90.4] weeks; Final analysis: 145.29 [3.3-225.3] weeks vs. 174.79 [0.9-226.1] weeks)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Placebo + Trastuzumab + Docetaxel | Arm B: Pertuzumab + Trastuzumab + Docetaxel
Number analyzed (Participants) | 121 | 122
months
  Primary Analysis | 12.4 [10.4 to 12.7] | 14.5 [12.5 to 18.6]
  Final Analysis | 12.5 [10.4 to 14.6] | 16.5 [12.7 to 20.2]
Statistical Analysis 1: Comparison: Arm A: Placebo + Trastuzumab + Docetaxel vs Arm B: Pertuzumab + Trastuzumab + Docetaxel; This was for the primary analysis. Hypothesis testing is considered exploratory in this bridging study; Test type: Other; p = 0.0418, Log Rank; A two-sided log-rank test was used, stratified by disease type and hormone-receptor status; Stratified Hazard Ratio = 0.69, 95% CI 2-sided [0.49 to 0.99] — This stratified Hazard Ratio (HR) is calculated as Arm B: Pertuzumab versus Arm A: Placebo. Cox proportional hazards model, stratified by disease type and hormone-receptor status, was used to estimate HR and its 95% CI
Statistical Analysis 2: Comparison: Arm A: Placebo + Trastuzumab + Docetaxel vs Arm B: Pertuzumab + Trastuzumab + Docetaxel; This was for the primary analysis. Hypothesis testing is considered exploratory in this bridging study; Test type: Other; p = 0.0556, Log Rank; This two-sided log-rank test was unstratified; Unstratified Hazard Ratio = 0.71, 95% CI 2-sided [0.50 to 1.01] — This unstratified Hazard Ratio (HR) is calculated as Arm B: Pertuzumab versus Arm A: Placebo. Cox proportional hazards model was used to estimate HR and its 95% CI
Statistical Analysis 3: Comparison: Arm A: Placebo + Trastuzumab + Docetaxel vs Arm B: Pertuzumab + Trastuzumab + Docetaxel; This was for the final analysis. Hypothesis testing is considered exploratory in this bridging study; Test type: Other; p = 0.0008, Log Rank; A two-sided log-rank test was used, stratified by disease type and hormone-receptor status; Stratified Hazard Ratio = 0.60, 95% CI 2-sided [0.45 to 0.81] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Arm A: Placebo + Trastuzumab + Docetaxel vs Arm B: Pertuzumab + Trastuzumab + Docetaxel; This was for the final analysis. Hypothesis testing is considered exploratory in this bridging study; Test type: Other; p = 0.0019, Log Rank; This two-sided log-rank test was unstratified; Unstratified Hazard Ratio = 0.63, 95% CI 2-sided [0.47 to 0.85] — [estimate comment as in outcome 1, analysis 2]

2. Primary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Event-Free for Progression-Free Survival at 1 to 3 Years, as Determined by the Investigator Using RECIST v1.1
Description: Progression-free survival (PFS) was defined as the time from randomization to first occurrence of progressive disease (PD), as determined by the investigator using RECIST v1.1, or death from any cause within 18 weeks after the last tumor assessment, whichever occurred first. As per RECIST v1.1, PD is a 20% increase in the sum of the diameters of target lesions, an increase in size of measurable lesions by at least 5 mm, and the appearance of new lesions. The Kaplan-Meier approach was used to estimate the percentage of participants who were event-free for PFS at 1, 2, and 3 years. Data for participants who did not have a PFS event were censored at the time of the last tumor assessment (if no tumor assessments performed after baseline visit, at randomization plus 1 day). At final analysis, the median [range] time on study for Arm A vs. Arm B was 145.29 [3.3-225.3] weeks vs. 174.79 [0.9-226.1] weeks.
Time Frame: At 1, 2, and 3 years
Population: ITT population: consists of all randomized participants, regardless of whether they received any study treatment. Participants are grouped according to the treatment group to which they were randomized. The number analyzed per timepoint represents the number of participants remaining at risk for a PFS event at that timepoint.
Measure: Number (95% Confidence Interval); unit: estimate of percentage of participants
Arm/Group | Arm A: Placebo + Trastuzumab + Docetaxel | Arm B: Pertuzumab + Trastuzumab + Docetaxel
Number analyzed (Participants) | 121 | 122
estimate of percentage of participants
  1 Year: number analyzed (Participants) | 59 | 77
  1 Year | 52.90 [43.75 to 62.04] | 66.37 [57.86 to 74.87]
  2 Years: number analyzed (Participants) | 21 | 42
  2 Years | 19.19 [11.85 to 26.53] | 37.85 [29.03 to 46.66]
  3 Years: number analyzed (Participants) | 13 | 29
  3 Years | 12.73 [6.48 to 18.97] | 29.44 [21.04 to 37.84]

3. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the time from randomization to death from any cause. The Kaplan-Meier approach was used to estimate median OS for each treatment arm. Participants who were alive or lost to follow-up at the time of the analysis were censored at the date they were last known to be alive. Participants with no post-baseline information were censored at the time of randomization plus 1 day. The results reported here are from the final analysis. At the primary completion date, the median duration of OS had not been reached and OS data was not considered mature due to the few number of events reported.
Time Frame: From date of randomization until the date of death from any cause (Median [range] time on study for Arm A vs. Arm B at Final analysis: 145.29 [3.3-225.3] weeks vs. 174.79 [0.9-226.1] weeks)
Population: ITT population: consists of all randomized participants, regardless of whether they received any study treatment. Participants are grouped according to the treatment group to which they were randomized.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Arm A: Placebo + Trastuzumab + Docetaxel | Arm B: Pertuzumab + Trastuzumab + Docetaxel
Number analyzed (Participants) | 121 | 122
months | NA [22.1 to NA] — The median duration of OS and the upper limit of the interquartile range were not estimable because too few events occurred during the study. | NA [30.6 to NA] — The median duration of OS and the upper limit of the interquartile range were not estimable because too few events occurred during the study.
Statistical Analysis 1: Comparison: Arm A: Placebo + Trastuzumab + Docetaxel vs Arm B: Pertuzumab + Trastuzumab + Docetaxel; Hypothesis testing is considered exploratory in this bridging study; Test type: Other; p = 0.0658, Log Rank; A two-sided log-rank test was used, stratified by disease type and hormone-receptor status; Stratified Hazard Ratio = 0.68, 95% CI 2-sided [0.45 to 1.03] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Arm A: Placebo + Trastuzumab + Docetaxel vs Arm B: Pertuzumab + Trastuzumab + Docetaxel; Hypothesis testing is considered exploratory in this bridging study; Test type: Other; p = 0.0864, Log Rank; This two-sided log-rank test was unstratified; Unstratified Hazard Ratio = 0.70, 95% CI 2-sided [0.46 to 1.06] — [estimate comment as in outcome 1, analysis 2]

4. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Event-Free for Overall Survival at 1 to 3 Years
Description: Overall survival (OS) was defined as the time from randomization to death from any cause. The Kaplan-Meier approach was used to estimate the percentage of participants who were event-free for OS (i.e., alive) at 1, 2, and 3 years. Participants who were alive or lost to follow-up at the time of the analysis were censored at the date they were last known to be alive. Participants with no post-baseline information were censored at the time of randomization plus 1 day. At final analysis, the median [range] time on study for Arm A vs. Arm B was 145.29 [3.3-225.3] weeks vs. 174.79 [0.9-226.1] weeks.
Time Frame: At 1, 2, and 3 Years
Population: ITT population: consists of all randomized participants, regardless of whether they received any study treatment. Participants are grouped according to the treatment group to which they were randomized. The number analyzed per timepoint represents the number of participants remaining at risk for an OS event at that timepoint.
Measure: Number (95% Confidence Interval); unit: estimate of percentage of participants
Arm/Group | Arm A: Placebo + Trastuzumab + Docetaxel | Arm B: Pertuzumab + Trastuzumab + Docetaxel
Number analyzed (Participants) | 121 | 122
estimate of percentage of participants
  1 Year: number analyzed (Participants) | 106 | 114
  1 Year | 90.64 [85.37 to 95.91] | 93.44 [89.05 to 97.84]
  2 Years: number analyzed (Participants) | 80 | 89
  2 Years | 73.85 [65.80 to 81.91] | 78.87 [71.50 to 86.24]
  3 Years: number analyzed (Participants) | 56 | 76
  3 Years | 58.41 [49.12 to 67.69] | 70.79 [62.50 to 79.09]

5. Secondary Outcome: Percentage of Participants With Measurable Disease at Baseline Who Achieved an Objective Response (Complete or Partial Response), as Determined by the Investigator Using RECIST v1.1
Description: An objective response was defined as a complete response (CR) or partial response (PR), as determined by the investigator using RECIST v1.1. As per RECIST v1.1, CR is defined as the disappearance of all target lesions, and PR is defined as at least a 30% decrease in the sum of diameters of target lesions. Also per RECIST v1.1, stable disease (SD) is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum on study; PD is defined as a 20% increase in the sum of the diameters of target lesions, an increase in size of measurable lesions by at least 5 mm, and the appearance of new lesions. The same assessment technique must be used throughout the study for evaluating a particular lesion, and the same investigator should assess all tumor responses for each participant. Participants without a post-baseline tumor assessment were considered non-responders.
Time Frame: At Baseline and every 9 weeks from date of randomization until disease progression or death, whichever occurs first (Median [range] time on study for Arm A vs. Arm B at Primary analysis: 57.14 [3.3-93.3] weeks vs. 59.64 [0.9-90.4] weeks)
Population: ITT population: consists of all randomized participants, regardless of whether they received any study treatment. Participants are grouped according to the treatment group to which they were randomized. Only participants with measurable disease at baseline were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Placebo + Trastuzumab + Docetaxel | Arm B: Pertuzumab + Trastuzumab + Docetaxel
Number analyzed (Participants) | 97 | 105
percentage of participants
  Objective Response (CR + PR) | 69.1 [58.88 to 78.07] | 79.0 [70.01 to 86.38]
  Complete Response (CR) | 8.2 [3.63 to 15.61] | 5.7 [2.13 to 12.02]
  Partial Response (PR) | 60.8 [50.39 to 70.58] | 73.3 [63.81 to 81.49]
  Stable Disease (SD) | 20.6 [13.07 to 30.03] | 15.2 [8.97 to 23.56]
  Progressive Disease (PD) | 4.1 [1.13 to 10.22] | 3.8 [1.05 to 9.47]
  Missing or Unevaluable | 6.2 [NA to NA] — 95% confidence intervals were only calculated for responses. | 1.9 [NA to NA] — 95% confidence intervals were only calculated for responses.
Statistical Analysis 1: Comparison: Arm A: Placebo + Trastuzumab + Docetaxel vs Arm B: Pertuzumab + Trastuzumab + Docetaxel; Hypothesis testing is considered exploratory in this bridging study; Test type: Other; p = 0.1126, Cochran-Mantel-Haenszel; Statistical test is stratified by disease type and hormone receptor status; Difference in Objective Response = 9.98, 95% CI 2-sided [-2.65 to 22.60] — The difference in objective response is calculated as Arm B: Pertuzumab minus Arm A: Placebo. 95% CI was calculated using Hauck-Anderson method
Statistical Analysis 2: Comparison: Arm A: Placebo + Trastuzumab + Docetaxel vs Arm B: Pertuzumab + Trastuzumab + Docetaxel; Hypothesis testing is considered exploratory in this bridging study; Test type: Other; p = 0.1108, Fisher Exact; Unadjusted; Difference in Objective Response = 9.98, 95% CI 2-sided [-2.65 to 22.60] — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: Duration of Objective Response, as Determined by the Investigator Using RECIST v1.1
Description: Duration of objective response was defined as the time from the first occurrence of a documented objective response (complete response [CR] or partial response [PR]) to the time of disease progression, as determined by the investigator using RECIST v1.1, or death from any cause within 18 weeks after the last tumor assessment, whichever occurred first. As per RECIST v1.1, CR is defined as the disappearance of all target lesions, and PR is defined as at least a 30% decrease in the sum of diameters of target lesions. The Kaplan-Meier approach was used to estimate median duration of objective response. Data for participants who did not have an event were censored at the time of the last tumor assessment (if no tumor assessments were performed after baseline visit, at randomization plus 1 day).
Time Frame: From date of first occurrence of documented objective response to date of event (Median [range] time on study for Arm A vs. Arm B at Primary analysis: 57.14 [3.3-93.3] weeks vs. 59.64 [0.9-90.4] weeks)
Population: ITT population: consists of all randomized participants, regardless of whether they received any study treatment. Participants are grouped according to the treatment group to which they were randomized. Only participants with measurable disease at baseline who achieved an objective response during the study were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Placebo + Trastuzumab + Docetaxel | Arm B: Pertuzumab + Trastuzumab + Docetaxel
Number analyzed (Participants) | 67 | 83
months | 10.4 [8.3 to 15.4] | 12.4 [10.6 to 14.9]
Statistical Analysis 1: Comparison: Arm A: Placebo + Trastuzumab + Docetaxel vs Arm B: Pertuzumab + Trastuzumab + Docetaxel; Hypothesis testing is considered exploratory in this bridging study; Test type: Other; p = 0.2867, Log Rank; Two-sided log-rank test was used, stratified by disease type and hormone-receptor status; Cox Proportional Hazard = 0.78, 95% CI 2-sided [0.49 to 1.24] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Number of Participants With at Least One Adverse Event
Description: The number of participants per treatment arm experiencing at least one adverse event, including all non-serious and serious adverse events, is reported here. Adverse events reported prior to first crossover treatment were included in the Placebo arm, and in the Crossover arm after that date, for participants in Arm A who crossed over from placebo to pertuzumab. At final analysis, the median [range] time on study treatment with placebo or pertuzumab per arm was: Arm A - Placebo: 52.3 [3-207] weeks; Arm B - Pertuzumab: 66.1 [3-225] weeks; Arm A - Crossover to Pertuzumab: 18.1 [12-24] weeks.
Time Frame: From first dose of study drug until 42 days after last dose of study drug (up to 4 years, 4 months)
Population: Safety population, which includes participants who received at least one dose of any study drug, with participants grouped according to the treatment received. Following approval of Protocol version 4 (07-March-2020), 12 Arm A participants who were receiving placebo crossed over to receive open-label treatment with pertuzumab.
Measure: Count of Participants; unit: Participants
Groups:
- Arm A: Crossover to Pertuzumab + Trastuzumab + Docetaxel: Following the primary analysis and upon approval of protocol version 4 (07-March-2020), the treatment assignment of participants in Arm A who were still on study treatment was unblinded, allowing the investigators to present those participants with the option to cross over and receive pertuzumab (in place of placebo) in addition to trastuzumab and docetaxel. Pertuzumab (840-mg loading dose for Cycle 1, followed by 420 mg for subsequent cycles), trastuzumab (8-mg/kg loading dose for Cycle 1, followed by 6 mg/kg for subsequent cycles), and docetaxel (75-mg/m^2) were administered by IV infusion every 3 weeks until disease progression or unacceptable toxicity.
Arm/Group | Arm A: Placebo + Trastuzumab + Docetaxel | Arm B: Pertuzumab + Trastuzumab + Docetaxel | Arm A: Crossover to Pertuzumab + Trastuzumab + Docetaxel
Number analyzed (Participants) | 120 | 122 | 12
Participants | 115 | 121 | 5

8. Secondary Outcome: Number of Participants With at Least One Grade ≥3 Adverse Event
Description: Adverse event (AE) severity was assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.0 (NCI-CTCAE v4.0); if the AE was not specifically listed, the following grades of severity were used: Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening or disabling; and Grade 5 = death. Severe and serious are not synonymous. Severity refers to the intensity of an AE, whereas a serious AE must meet criteria set out in the protocol; both were independently assessed for each AE. AEs reported prior to first crossover treatment were included in the Placebo arm, and in the Crossover arm after that date, for participants in Arm A who crossed over from placebo to pertuzumab. At final analysis, the median [range] time on study treatment with placebo or pertuzumab per arm was: Arm A - Placebo: 52.3 [3-207] weeks; Arm B - Pertuzumab: 66.1 [3-225] weeks; Arm A - Crossover to Pertuzumab: 18.1 [12-24] weeks.
Time Frame: From first dose of study drug until 42 days after last dose of study drug (up to 4 years, 4 months)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Placebo + Trastuzumab + Docetaxel | Arm B: Pertuzumab + Trastuzumab + Docetaxel | Arm A: Crossover to Pertuzumab + Trastuzumab + Docetaxel
Number analyzed (Participants) | 120 | 122 | 12
Participants | 83 | 90 | 1

9. Secondary Outcome: Number of Participants With at Least One Adverse Event Leading to Withdrawal From Any Treatment
Description: Adverse events reported prior to first crossover treatment were included in the Placebo arm, and in the Crossover arm after that date, for participants in Arm A who crossed over from placebo to pertuzumab. At final analysis, the median [range] time on study treatment with placebo or pertuzumab per arm was: Arm A - Placebo: 52.3 [3-207] weeks; Arm B - Pertuzumab: 66.1 [3-225] weeks; Arm A - Crossover to Pertuzumab: 18.1 [12-24] weeks.
Time Frame: From first dose of study drug until 42 days after last dose of study drug (up to 4 years, 4 months)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Placebo + Trastuzumab + Docetaxel | Arm B: Pertuzumab + Trastuzumab + Docetaxel | Arm A: Crossover to Pertuzumab + Trastuzumab + Docetaxel
Number analyzed (Participants) | 120 | 122 | 12
Participants | 10 | 15 | 0

10. Secondary Outcome: Number of Participants With Symptomatic Left Ventricular Systolic Dysfunction (LVSD), as Determined Using Echocardiography (ECHO) or Multiple-Gated Acquisition (MUGA) Scan
Description: The number of participants with symptomatic left ventricular systolic dysfunction (LVSD) at any time during the study, as determined using echocardiography (ECHO) or multiple-gated acquisition (MUGA) scan, were summarized by treatment arm. Symptomatic LVSD was evaluated according to NCI CTCAE v4.0 (for "heart failure") and the New York Heart Association (NYHA) classification. At final analysis, the median [range] time on study treatment with placebo or pertuzumab per arm was: Arm A - Placebo: 52.3 [3-207] weeks; Arm B - Pertuzumab: 66.1 [3-225] weeks; Arm A - Crossover to Pertuzumab: 18.1 [12-24] weeks.
Time Frame: From first dose of study drug until 42 days after last dose of study drug (up to 4 years, 4 months)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Placebo + Trastuzumab + Docetaxel | Arm B: Pertuzumab + Trastuzumab + Docetaxel | Arm A: Crossover to Pertuzumab + Trastuzumab + Docetaxel
Number analyzed (Participants) | 120 | 122 | 12
Participants | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With an Asymptomatic Decline in Left Ventricular Ejection Fraction (LVEF) Event, as Determined Using ECHO or MUGA Scan
Description: An asymptomatic decline in LVEF event is reported as an adverse event of "ejection fraction decreased" and is defined as either of the following: an absolute decrease in LVEF of ≥10 percentage points from baseline to an LVEF of <50%; or an asymptomatic decrease in LVEF requiring treatment or leading to discontinuation of pertuzumab (or placebo) and trastuzumab. At final analysis, the median [range] time on study treatment with placebo or pertuzumab per arm was: Arm A - Placebo: 52.3 [3-207] weeks; Arm B - Pertuzumab: 66.1 [3-225] weeks; Arm A - Crossover to Pertuzumab: 18.1 [12-24] weeks.
Time Frame: From first dose of study drug until 42 days after last dose of study drug (up to 4 years, 4 months)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Placebo + Trastuzumab + Docetaxel | Arm B: Pertuzumab + Trastuzumab + Docetaxel | Arm A: Crossover to Pertuzumab + Trastuzumab + Docetaxel
Number analyzed (Participants) | 120 | 122 | 12
Participants | 0 | 2 | 0

12. Secondary Outcome: Number of Participants by the LVEF Abnormality Status Categories Over Time, as Determined by the Change From Baseline in LVEF Using ECHO or MUGA Scans
Description: Left ventricular ejection fraction (LVEF) is the measurement of how much blood is being pumped out of the left ventricle of the heart with each contraction. LVEF was calculated using the modified Simpson method and must have been ≥55% at baseline as determined by the local facility before a participant could be enrolled in the study. The investigator decided which method of LVEF assessment (ECHO [preferred] or MUGA scan) would be used for each participant at baseline, and the same method was to be used throughout the study, to the extent possible. The LVEF abnormality status categories, as a change relative to LVEF at baseline, included: Increase or no change in LVEF; Decrease of <10 LVEF points; Absolute LVEF value ≥50% and a decrease of ≥10 LVEF points; and Absolute LVEF value <50% and a decrease of ≥10 LVEF points. The overall worst LVEF value was defined as the lowest post-baseline value up to the end of the study, including unscheduled assessments and the post-treatment period.
Time Frame: Baseline, Weeks 9, 18, 27, 36, 45, 54, 63, 72, 81, 90, 99, 108, 117, 126, 135, 144, 153, 162, 171, 180, 189, 198, 207, 216, and 225, Study Drug Discontinuation Visit (up to 4 years, 4 months), and Treatment-Free Follow-Up at 6 months, and 1 and 2 years
Population: Safety population, which includes participants who received at least one dose of any study drug, with participants grouped according to the treatment received. Number analyzed indicates the number of participants with a baseline LVEF measurement and a post-baseline LVEF measurement at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Placebo + Trastuzumab + Docetaxel | Arm B: Pertuzumab + Trastuzumab + Docetaxel
Number analyzed (Participants) | 120 | 122
Participants
  Week 9: number analyzed (Participants) | 111 | 119
  Week 9: Increase or No Change in LVEF | 57 | 63
  Week 9: Decrease <10 LVEF Points | 51 | 52
  Week 9: Absolute Value ≥50% & Decrease ≥10 LVEF Points | 3 | 4
  Week 9: Absolute Value <50% & Decrease ≥10 LVEF Points | 0 | 0
  Week 18: number analyzed (Participants) | 98 | 111
  Week 18: Increase or No Change in LVEF | 61 | 62
  Week 18: Decrease <10 LVEF Points | 33 | 45
  Week 18: Absolute Value ≥50% & Decrease ≥10 LVEF Points | 4 | 3
  Week 18: Absolute Value <50% & Decrease ≥10 LVEF Points | 0 | 1
  Week 27: number analyzed (Participants) | 92 | 99
  Week 27: Increase or No Change in LVEF | 54 | 51
  Week 27: Decrease <10 LVEF Points | 35 | 43
  Week 27: Absolute Value ≥50% & Decrease ≥10 LVEF Points | 3 | 5
  Week 27: Absolute Value <50% & Decrease ≥10 LVEF Points | 0 | 0
  Week 36: number analyzed (Participants) | 76 | 94
  Week 36: Increase or No Change in LVEF | 45 | 46
  Week 36: Decrease <10 LVEF Points | 28 | 43
  Week 36: Absolute Value ≥50% & Decrease ≥10 LVEF Points | 3 | 4
  Week 36: Absolute Value <50% & Decrease ≥10 LVEF Points | 0 | 1
  Week 45: number analyzed (Participants) | 68 | 82
  Week 45: Increase or No Change in LVEF | 34 | 36
  Week 45: Decrease <10 LVEF Points | 29 | 43
  Week 45: Absolute Value ≥50% & Decrease ≥10 LVEF Points | 5 | 3
  Week 45: Absolute Value <50% & Decrease ≥10 LVEF Points | 0 | 0
  Week 54: number analyzed (Participants) | 57 | 75
  Week 54: Increase or No Change in LVEF | 26 | 38
  Week 54: Decrease <10 LVEF Points | 27 | 34
  Week 54: Absolute Value ≥50% & Decrease ≥10 LVEF Points | 4 | 3
  Week 54: Absolute Value <50% & Decrease ≥10 LVEF Points | 0 | 0
  Week 63: number analyzed (Participants) | 44 | 66
  Week 63: Increase or No Change in LVEF | 21 | 30
  Week 63: Decrease <10 LVEF Points | 17 | 33
  Week 63: Absolute Value ≥50% & Decrease ≥10 LVEF Points | 6 | 3
  Week 63: Absolute Value <50% & Decrease ≥10 LVEF Points | 0 | 0
  Week 72: number analyzed (Participants) | 37 | 61
  Week 72: Increase or No Change in LVEF | 17 | 26
  Week 72: Decrease <10 LVEF Points | 15 | 31
  Week 72: Absolute Value ≥50% & Decrease ≥10 LVEF Points | 5 | 4
  Week 72: Absolute Value <50% & Decrease ≥10 LVEF Points | 0 | 0
  Week 81: number analyzed (Participants) | 34 | 55
  Week 81: Increase or No Change in LVEF | 19 | 29
  Week 81: Decrease <10 LVEF Points | 12 | 24
  Week 81: Absolute Value ≥50% & Decrease ≥10 LVEF Points | 3 | 2
  Week 81: Absolute Value <50% & Decrease ≥10 LVEF Points | 0 | 0
  Week 90: number analyzed (Participants) | 30 | 47
  Week 90: Increase or No Change in LVEF | 17 | 24
  Week 90: Decrease <10 LVEF Points | 11 | 20
  Week 90: Absolute Value ≥50% & Decrease ≥10 LVEF Points | 2 | 3
  Week 90: Absolute Value <50% & Decrease ≥10 LVEF Points | 0 | 0
  Week 99: number analyzed (Participants) | 26 | 46
  Week 99: Increase or No Change in LVEF | 14 | 21
  Week 99: Decrease <10 LVEF Points | 10 | 23
  Week 99: Absolute Value ≥50% & Decrease ≥10 LVEF Points | 2 | 2
  Week 99: Absolute Value <50% & Decrease ≥10 LVEF Points | 0 | 0
  Week 108: number analyzed (Participants) | 21 | 42
  Week 108: Increase or No Change in LVEF | 13 | 15
  Week 108: Decrease <10 LVEF Points | 7 | 24
  Week 108: Absolute Value ≥50% & Decrease ≥10 LVEF Points | 1 | 3
  Week 108: Absolute Value <50% & Decrease ≥10 LVEF Points | 0 | 0
  Week 117: number analyzed (Participants) | 18 | 39
  Week 117: Increase or No Change in LVEF | 14 | 18
  Week 117: Decrease <10 LVEF Points | 3 | 18
  Week 117: Absolute Value ≥50% & Decrease ≥10 LVEF Points | 1 | 3
  Week 117: Absolute Value <50% & Decrease ≥10 LVEF Points | 0 | 0
  Week 126: number analyzed (Participants) | 17 | 37
  Week 126: Increase or No Change in LVEF | 7 | 20
  Week 126: Decrease <10 LVEF Points | 9 | 15
  Week 126: Absolute Value ≥50% & Decrease ≥10 LVEF Points | 1 | 2
  Week 126: Absolute Value <50% & Decrease ≥10 LVEF Points | 0 | 0
  Week 135: number analyzed (Participants) | 15 | 35
  Week 135: Increase or No Change in LVEF | 6 | 15
  Week 135: Decrease <10 LVEF Points | 8 | 18
  Week 135: Absolute Value ≥50% & Decrease ≥10 LVEF Points | 1 | 2
  Week 135: Absolute Value <50% & Decrease ≥10 LVEF Points | 0 | 0
  Week 144: number analyzed (Participants) | 14 | 31
  Week 144: Increase or No Change in LVEF | 10 | 18
  Week 144: Decrease <10 LVEF Points | 3 | 10
  Week 144: Absolute Value ≥50% & Decrease ≥10 LVEF Points | 1 | 3
  Week 144: Absolute Value <50% & Decrease ≥10 LVEF Points | 0 | 0
  Week 153: number analyzed (Participants) | 14 | 30
  Week 153: Increase or No Change in LVEF | 7 | 12
  Week 153: Decrease <10 LVEF Points | 7 | 15
  Week 153: Absolute Value ≥50% & Decrease ≥10 LVEF Points | 0 | 3
  Week 153: Absolute Value <50% & Decrease ≥10 LVEF Points | 0 | 0
  Week 162: number analyzed (Participants) | 13 | 30
  Week 162: Increase or No Change in LVEF | 7 | 17
  Week 162: Decrease <10 LVEF Points | 6 | 12
  Week 162: Absolute Value ≥50% & Decrease ≥10 LVEF Points | 0 | 1
  Week 162: Absolute Value <50% & Decrease ≥10 LVEF Points | 0 | 0
  Week 171: number analyzed (Participants) | 12 | 28
  Week 171: Increase or No Change in LVEF | 7 | 10
  Week 171: Decrease <10 LVEF Points | 4 | 16
  Week 171: Absolute Value ≥50% & Decrease ≥10 LVEF Points | 1 | 2
  Week 171: Absolute Value <50% & Decrease ≥10 LVEF Points | 0 | 0
  Week 180: number analyzed (Participants) | 12 | 23
  Week 180: Increase or No Change in LVEF | 9 | 8
  Week 180: Decrease <10 LVEF Points | 3 | 14
  Week 180: Absolute Value ≥50% & Decrease ≥10 LVEF Points | 0 | 1
  Week 180: Absolute Value <50% & Decrease ≥10 LVEF Points | 0 | 0
  Week 189: number analyzed (Participants) | 9 | 15
  Week 189: Increase or No Change in LVEF | 5 | 6
  Week 189: Decrease <10 LVEF Points | 3 | 9
  Week 189: Absolute Value ≥50% & Decrease ≥10 LVEF Points | 1 | 0
  Week 189: Absolute Value <50% & Decrease ≥10 LVEF Points | 0 | 0
  Week 198: number analyzed (Participants) | 7 | 11
  Week 198: Increase or No Change in LVEF | 4 | 6
  Week 198: Decrease <10 LVEF Points | 2 | 5
  Week 198: Absolute Value ≥50% & Decrease ≥10 LVEF Points | 1 | 0
  Week 198: Absolute Value <50% & Decrease ≥10 LVEF Points | 0 | 0
  Week 207: number analyzed (Participants) | 3 | 8
  Week 207: Increase or No Change in LVEF | 2 | 5
  Week 207: Decrease <10 LVEF Points | 1 | 3
  Week 207: Absolute Value ≥50% & Decrease ≥10 LVEF Points | 0 | 0
  Week 207: Absolute Value <50% & Decrease ≥10 LVEF Points | 0 | 0
  Week 216: number analyzed (Participants) | 1 | 4
  Week 216: Increase or No Change in LVEF | 1 | 3
  Week 216: Decrease <10 LVEF Points | 0 | 1
  Week 216: Absolute Value ≥50% & Decrease ≥10 LVEF Points | 0 | 0
  Week 216: Absolute Value <50% & Decrease ≥10 LVEF Points | 0 | 0
  Week 225: number analyzed (Participants) | 0 | 1
  Week 225: Increase or No Change in LVEF |  | 1
  Week 225: Decrease <10 LVEF Points |  | 0
  Week 225: Absolute Value ≥50% & Decrease ≥10 LVEF Points |  | 0
  Week 225: Absolute Value <50% & Decrease ≥10 LVEF Points |  | 0
  Study Drug Discontinuation Visit: number analyzed (Participants) | 81 | 87
  Study Drug Discontinuation Visit: Increase or No Change in LVEF | 45 | 45
  Study Drug Discontinuation Visit: Decrease <10 LVEF Points | 28 | 39
  Study Drug Discontinuation Visit: Absolute Value ≥50% & Decrease ≥10 LVEF Points | 8 | 3
  Study Drug Discontinuation Visit: Absolute Value <50% & Decrease ≥10 LVEF Points | 0 | 0
  Treatment-Free Follow-Up at 6 Months: number analyzed (Participants) | 43 | 36
  Treatment-Free Follow-Up at 6 Months: Increase or No Change in LVEF | 20 | 18
  Treatment-Free Follow-Up at 6 Months: Decrease <10 LVEF Points | 20 | 18
  Treatment-Free Follow-Up at 6 Months: Absolute Value ≥50% & Decrease ≥10 LVEF Points | 3 | 0
  Treatment-Free Follow-Up at 6 Months: Absolute Value <50% & Decrease ≥10 LVEF Points | 0 | 0
  Treatment-Free Follow-Up at 1 Year: number analyzed (Participants) | 23 | 19
  Treatment-Free Follow-Up at 1 Year: Increase or No Change in LVEF | 13 | 4
  Treatment-Free Follow-Up at 1 Year: Decrease <10 LVEF Points | 10 | 14
  Treatment-Free Follow-Up at 1 Year: Absolute Value ≥50% & Decrease ≥10 LVEF Points | 0 | 1
  Treatment-Free Follow-Up at 1 Year: Absolute Value <50% & Decrease ≥10 LVEF Points | 0 | 0
  Treatment-Free Follow-Up at 2 Years: number analyzed (Participants) | 3 | 4
  Treatment-Free Follow-Up at 2 Years: Increase or No Change in LVEF | 1 | 2
  Treatment-Free Follow-Up at 2 Years: Decrease <10 LVEF Points | 0 | 1
  Treatment-Free Follow-Up at 2 Years: Absolute Value ≥50% & Decrease ≥10 LVEF Points | 2 | 1
  Treatment-Free Follow-Up at 2 Years: Absolute Value <50% & Decrease ≥10 LVEF Points | 0 | 0
  Overall Worst LVEF Value (Maximum LVEF Decrease): number analyzed (Participants) | 112 | 119
  Overall Worst LVEF Value (Maximum LVEF Decrease): Increase or No Change in LVEF | 21 | 20
  Overall Worst LVEF Value (Maximum LVEF Decrease): Decrease <10 LVEF Points | 75 | 75
  Overall Worst LVEF Value (Maximum LVEF Decrease): Absolute Value ≥50% & Decrease ≥10 LVEF Points | 16 | 22
  Overall Worst LVEF Value (Maximum LVEF Decrease): Absolute Value <50% & Decrease ≥10 LVEF Points | 0 | 2

13. Secondary Outcome: Baseline LVEF and Change From Baseline to Maximum On-Treatment Decrease in LVEF at Any Point During the Study
Description: The baseline left ventricular ejection fraction (LVEF) and change from baseline to the maximum on-treatment decrease in LVEF at any point during the study are reported here. LVEF is the measurement of how much blood is being pumped out of the left ventricle of the heart (the main pumping chamber) with each contraction. LVEF was calculated using the modified Simpson method and must have been ≥55% at baseline as determined by the local facility before a participant could be enrolled in the study. The investigator decided which method of LVEF assessment (ECHO [preferred] or MUGA scan) would be used for each participant at baseline, and the same method should have been used throughout the study, to the extent possible. At final analysis, the median [range] time on study for Arm A vs. Arm B was 145.29 [3.3-225.3] weeks vs. 174.79 [0.9-226.1] weeks.
Time Frame: Baseline and every 9 weeks from date of randomization until treatment discontinuation (up to 4 years, 4 months)
Population: Safety population, which includes participants who received at least one dose of any study drug, with participants grouped according to the treatment received. Number analyzed indicates participants with a baseline LVEF measurement and at least one post-baseline LVEF measurement, respectively.
Measure: Mean (Standard Deviation); unit: percentage points of LVEF
Arm/Group | Arm A: Placebo + Trastuzumab + Docetaxel | Arm B: Pertuzumab + Trastuzumab + Docetaxel
Number analyzed (Participants) | 120 | 122
percentage points of LVEF
  Baseline LVEF (value at visit): number analyzed (Participants) | 119 | 122
  Baseline LVEF (value at visit) | 64.23 (4.90) | 65.08 (4.43)
  Change from Baseline to Max Decrease in LVEF: number analyzed (Participants) | 112 | 119
  Change from Baseline to Max Decrease in LVEF | -4.88 (5.41) | -5.48 (5.06)
Statistical Analysis 1: Comparison: Arm A: Placebo + Trastuzumab + Docetaxel vs Arm B: Pertuzumab + Trastuzumab + Docetaxel; Test type: Other; Mean Difference (Net) = -0.60, 95% CI 2-sided [-1.96 to 0.75] — The treatment difference for change from baseline to maximum on-treatment decrease in LVEF is defined as Arm B: Pertuzumab minus Arm A: Placebo

ADVERSE EVENTS:
Time Frame: From first dose of study drug until 42 days after last dose of study drug (up to 4 years, 4 months). At final analysis, the median [range] time on study treatment with placebo or pertuzumab per arm was: Arm A - Placebo: 52.3 [3-207] weeks; Arm B - Pertuzumab: 66.1 [3-225] weeks; Arm A - Crossover to Pertuzumab: 18.1 [12-24] weeks.
Arm/Group | Arm A: Placebo + Trastuzumab + Docetaxel | Arm B: Pertuzumab + Trastuzumab + Docetaxel | Arm A: Crossover to Pertuzumab + Trastuzumab + Docetaxel
All-Cause Mortality (participants affected / at risk) | 50/120 | 40/122 | 0/12
Serious Adverse Events (participants affected / at risk) | 23/120 | 30/122 | 1/12
Other Adverse Events (participants affected / at risk) | 114/120 | 119/122 | 5/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Placebo + Trastuzumab + Docetaxel (N=120) | Arm B: Pertuzumab + Trastuzumab + Docetaxel (N=122) | Arm A: Crossover to Pertuzumab + Trastuzumab + Docetaxel (N=12)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 3 (3) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (3) | 3 (3) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 8 (16) | 9 (16) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1) | 0 (0)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 5 (5) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Placebo + Trastuzumab + Docetaxel (N=120) | Arm B: Pertuzumab + Trastuzumab + Docetaxel (N=122) | Arm A: Crossover to Pertuzumab + Trastuzumab + Docetaxel (N=12)
Anaemia (Blood and lymphatic system disorders) | 58 (112) | 67 (179) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 87 (319) | 91 (349) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 81 (305) | 87 (314) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 12 (28) | 9 (25) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 6 (6) | 7 (11) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 8 (13) | 8 (9) | 0 (0)
Constipation (Gastrointestinal disorders) | 11 (15) | 8 (10) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 28 (57) | 56 (102) | 0 (0)
Flatulence (Gastrointestinal disorders) | 4 (5) | 8 (8) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 6 (7) | 10 (16) | 0 (0)
Nausea (Gastrointestinal disorders) | 15 (24) | 15 (28) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 4 (6) | 15 (20) | 0 (0)
Vomiting (Gastrointestinal disorders) | 11 (13) | 13 (28) | 0 (0)
Asthenia (General disorders) | 20 (45) | 25 (38) | 0 (0)
Fatigue (General disorders) | 7 (10) | 5 (5) | 0 (0)
Influenza like illness (General disorders) | 6 (7) | 9 (13) | 0 (0)
Malaise (General disorders) | 11 (14) | 9 (16) | 0 (0)
Oedema peripheral (General disorders) | 18 (31) | 12 (17) | 0 (0)
Pain (General disorders) | 22 (30) | 19 (39) | 0 (0)
Pyrexia (General disorders) | 21 (28) | 29 (46) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 6 (8) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 7 (8) | 9 (14) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 16 (18) | 17 (20) | 0 (0)
Alanine aminotransferase increased (Investigations) | 56 (101) | 45 (83) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 49 (98) | 45 (95) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 9 (13) | 9 (14) | 1 (2)
Blood bilirubin increased (Investigations) | 14 (28) | 14 (20) | 0 (0)
Blood creatinine increased (Investigations) | 8 (10) | 11 (26) | 1 (1)
Blood triglycerides increased (Investigations) | 4 (13) | 7 (16) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 10 (12) | 8 (11) | 0 (0)
Weight decreased (Investigations) | 6 (8) | 11 (12) | 0 (0)
Weight increased (Investigations) | 16 (20) | 4 (5) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 14 (19) | 15 (15) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 8 (9) | 14 (25) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8 (10) | 11 (17) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 8 (24) | 18 (45) | 1 (1)
Hypoproteinaemia (Metabolism and nutrition disorders) | 3 (3) | 7 (7) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 7 (10) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 7 (8) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (13) | 4 (4) | 0 (0)
Dizziness (Nervous system disorders) | 11 (13) | 7 (8) | 0 (0)
Headache (Nervous system disorders) | 8 (11) | 9 (11) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 8 (9) | 13 (13) | 0 (0)
Neurotoxicity (Nervous system disorders) | 7 (7) | 9 (10) | 0 (0)
Insomnia (Psychiatric disorders) | 10 (12) | 10 (17) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (21) | 26 (33) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (11) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 40 (40) | 50 (53) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 (4) | 7 (8) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 15 (15) | 12 (12) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (7) | 8 (13) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 11 (13) | 11 (22) | 0 (0)
Hypertension (Vascular disorders) | 8 (10) | 12 (15) | 0 (0)
Palpitations (Cardiac disorders) | 8 (16) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 6 (9) | 6 (8) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (5) | 8 (10) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-03-07): https://cdn.clinicaltrials.gov/large-docs/55/NCT02896855/Prot_002.pdf
  • Statistical Analysis Plan (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/55/NCT02896855/SAP_001.pdf